CLINICAL TRIAL: NCT05803070
Title: Topical Cetirizine Versus Topical Betamethasone in Treatment of Localized Alopecia Areata
Brief Title: Topical Cetirizine in Treatment of Localized Alopecia Areata
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Esam Fathy, doctor, Assiut University
Other Study IDs: Alopecia areata treatment
Record Dates: First submitted 2023-03-15; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Alopecia Areata
Keywords: Cetirizine
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: patients with alopecia areata who will be treated with topical cetirizine 1%
  Interventions: Drug: Topical Cetirizine 1 %
- B: patients with alopecia areata who will be treated with topical betamethasone valerate 0.1%
  Interventions: Drug: Topical betamethasone valerate 0.1%

INTERVENTIONS:
Drug: Topical Cetirizine 1 % — topical cetirizine belongs to anti histamines group
  Groups: A
Drug: Topical betamethasone valerate 0.1% — topical betamethasone valerate belongs to corticosteroids group
  Groups: B

SUMMARY:
Evaluate and compare the efficacy and safety of topical cetirizine 1%, versus topical betamethasone valerate 0.1% in the treatment of localized alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata (AA) is one of the commonest autoimmune non-cicatricial hair loss that affects different parts of hair-bearing areas of the body . Nearly 2% of the population at some stage of their life may be affected by alopecia areata while the prevalence of alopecia areata was reported to be between 0.1% to 0.2%. Alopecia areata can occur at any age, although it starts in the first three decades of life in most patients, and both sexes are equally affected. It can present clinically as a well-defined patch of hair loss, diffuse hair loss, reticulate hair loss, ophiasis, ophiasis inversus, alopecia totalis (complete loss of scalp hair), or alopecia universalis (hair loss of all over the body).

Many treatment options including topical, systemic, injectable and laser modalities have been used for the treatment of AA . Among the various treatment options for alopecia areata, topical corticosteroids as betamethasone valerate are considered as standard therapy.

There have been reports on the efficacy/adjunctive role of systemic antihistamines in alopecia areata. Moreover, fexofenadine was found to enhance hair regrowth in two cases of extensive resistant alopecia areata.

Cetirizine hydrochloride belongs to a family of medicines called antihistamines which has varied medical uses and is commonly used to relieve allergy symptoms such as watery eyes, runny nose, sneezing, hives, and itching. In addition, it has been demonstrated that cetirizine inhibits release of prostaglandin D2 and stimulates the release of prostaglandin E2 .

Topical cetirizine was used with good results and with no notable side effects for the treatment of androgenic alopecia. Because of this evidence and the absence of hormonal influence, cetirizine was considered suitable for this kind of hair loss .

Cetirizine is able to increase prostaglandins (PG) E and Fα synthesis, and thus, reduce inflammation. It also decreases prostaglandin D2 (PGD2) synthesis. Prostaglandins E and Fα influence positively hair follicle growth, and stimulate and maintain the anagen phase. So, by increasing the synthesis of prostaglandins E and Fα, cetirizine induces an increase in total and terminal hair density and hair diameter, and a reduction in vellus hair density.

A recent study has shown a significantly increased expression of prostaglandin D2 in the serum and lesional skin of alopecia areata patients than in controls. Also, a case report has demonstrated the improvement of diffuse alopecia caused by palbociclib for the treatment of breast cancer, using topical cetirizine 0.5% solution.

Dermoscopy is a non-invasive diagnostic utility, used to evaluate many skin and hair disorders. It may aid in the diagnosis of many uncertain hair disorders, one of which is alopecia areata. Different dermoscopic characteristics are seen in alopecia areata such as, black dots, yellow dots, tapering hairs (exclamation mark hairs). broken hairs and short vellus hairs.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sex with age ≥ 12 years.
* Localized alopecia areata: <50% affection of the scalp surface.
* Stable disease (no new patches or increase in size for at least 2 weeks)

Exclusion Criteria:

* Uncertain diagnosis.
* Age < 12 years.
* Severe forms of alopecia (extensive alopecia; > 50% of scalp surface), ophiasis type, alopecia totalis or alopecia universalis.
* Alopecia Areata outside the scalp.
* Patients who have received topical treatment for alopecia areata in the past month.
* Patients who have received systemic treatment for alopecia areata in the past 2 months.
* Any associated skin or hair disorders.
* Any associated medical condition requiring oral corticosteroids, immunosuppressive or light therapy.
* Presence of any systemic autoimmune disease.
* Pregnant and lactating women
* Unrealistic expectations.

Ages: 12 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with alopecia areata who attend the outpatient clinic of Dematology department ,Assuit University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Compare topical cetirizine and betamethasone valerate in treatment of alopecia areata | baseline
  compare the healing rate
Clinical evaluation by SALT score | baseline
  an ideal objective method of follow-up and good evaluation of any therapeutic option
Clinical evaluation by photographic evaluation | baseline
  The photographs and response to treatment will be evaluated objectively by two-blinded dermatologists using a five-point semiquantitative score (regrowth scale) defined as follows: 0 score (regrowth <10%), 1 score (regrowth 11-25%), 2 score (regrowth 26-50%), 3 score (regrowth 51-75%), 4 score (≥ 75)
Clinical evaluation by patient's satisfaction level | baseline
  Asking the patients about their satisfaction towards treatment using a five-point scale (-1: condition worsened, 0: not satisfied, 1: poorly satisfied, 2: moderately satisfied, 3: very satisfied)

REFERENCES:
- [Background] Rossi A, Campo D, Fortuna MC, Garelli V, Pranteda G, De Vita G, Sorriso-Valvo L, Di Nunno D, Carlesimo M. A preliminary study on topical cetirizine in the therapeutic management of androgenetic alopecia. J Dermatolog Treat. 2018 Mar;29(2):149-151. doi: 10.1080/09546634.2017.1341610. Epub 2017 Jun 29. PMID 28604133